CLINICAL TRIAL: NCT05619926
Title: A Multi-center, Open-label, Multiple-dose Design, Phase 2 Trial to Evaluate the Safety and Efficacy of STSP-0601 for Injection in Patients With Hemophilia Without Inhibitor
Brief Title: Safety and Efficacy of STSP-0601 in Adult Patients With Hemophilia A or B Without Inhibitor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Staidson (Beijing) Biopharmaceuticals Co., Ltd (Industry)
Collaborators: Beijing Novikang Medical Technology Co., LTD (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STSP-0601-03
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-08

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Consecutive doses of low-dose of STSP-0601 (Experimental)
  Interventions: Drug: STSP-0601 for Injection
- Consecutive doses of high-dose of STSP-0601 (Experimental)
  Interventions: Drug: STSP-0601 for Injection

INTERVENTIONS:
Drug: STSP-0601 for Injection — Intravenous Injection

SUMMARY:
This study will assess the safety,efficacy,pharmacokinetics and pharmacodynamics of multiple-dose of STSP-0601 at two dose levels for the treatment of bleeding episodes in hemophilia A or B patients without inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* 18 ≤age≤70 years of age,male;
* Hemophilia A or B patients;
* A bleeding event requiring treatment occurred (Only applicable to the on-demand treatment stage);
* Factor VIII or IX level <2%, inhibitor titer < 0.6 BU;
* There were at least 2 bleeding events that requiring treatment occurred in the past 6 months before screening (Only the second stage is applicable);
* Establish proper venous access;
* Agree to use adequate contraception to avoid pregnancy;
* Provide signed informed consent.

Exclusion Criteria:

* Have any coagulation disorder other than hemophilia;
* Plan to receive prophylactic treatment of coagulation factor during the trail;
* 4 weeks before screening, receive prophylactic treatment of amesetuzumab or plan to receive prophylactic treatment of amesetuzumab during the trial;
* Patients received anticoagulant or antifibrinolytic therapy 7 days before enrollment or plan to receive these drugs during the trial;
* Patients received anticoagulation therapy (such as coagulation factor replacement therapy, prothrombin complex, plasma, etc.) 7 days before enrollment;
* Have a history of arterial and/or venous thrombotic events;
* Platelet <100×109/L;
* Hemoglobin<90g/L;
* Severe liver or kidney disease;
* Severe bleeding event occurred within 4 weeks before enrollment;
* Accepted major operation or blood transfusion within 4 weeks before enrollment;
* HIV positive;
* Have a known allergy to STSP-0601;
* Participate in other clinical research within 4 weeks before enrollment(except for participating in prothrombin complex, FVII, FVIIa, FVIII, FIX trails);
* Patients not suitable for the trail according to the judgment of the investigators.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | From day 0 to up to day 4
Proportion of successfully treated bleeding episodes | 8 hours after first administration of study drug

SECONDARY OUTCOMES:
Proportion of successfully treated bleeding episodes | 12 hours，24 hours after first administration of study drug
Proportion of bleeding episodes received salvage treatment | Within 3 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Principal Investigator — Affiliation:Hospital of Hematology, Chinese Academy of Medical Sciences
Locations (12):
- China (12):
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Lanzhou University First Hospita, Lanzhou, Gansu
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - North China University of Technology Affiliated Hospital, Tangshan, Hebei
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing Gulou Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Xi'an Central Hospital, Xi’an, Shanxi
  - Hospital of Hematology, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No